CLINICAL TRIAL: NCT06550362
Title: A Randomized Controlled Trial Comparing Daily Oral Iron Administration to Every Alternate Day Iron Administration in the Treatment of Iron Deficiency Anemia in Pediatric Patients.
Brief Title: Daily Iron vs Every-other-day Iron for Pediatric Patients With IDA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5240248
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Iron every other day (Experimental): Oral iron daily at 6 mg (elemental)/kg/day (max 200 mg elemental) taken every other day.
  Interventions: Drug: iron sulfate
- Iron every day (Active Comparator): Oral iron daily at 6 mg (elemental)/kg/day (max 200 mg elemental) taken every day.
  Interventions: Drug: iron sulfate

INTERVENTIONS:
Drug: iron sulfate — Oral iron administration

SUMMARY:
Iron Deficiency Anemia (IDA) is a prevalent global health issue affecting a significant proportion of the population, including children. While daily oral iron supplementation is a common approach to treat IDA, concerns regarding side effects and compliance have led to exploration of alternative dosing schedules, such as every-other-day. This study aims to investigate the efficacy and safety of daily versus every other day oral iron supplementation in the management of IDA in pediatric patients.

DETAILED DESCRIPTION:
This is a prospective open-label randomized controlled study. Patients will be randomized into two groups, one group (investigational) will receive oral iron every other day (every 48 hours) and the control group will be prescribed daily oral iron. Data will be collected prospectively including compliance assessment, side effect profile, hemoglobin (CBC), iron stores, hepcidin levels and other monitoring as relevant for best patient care.

At the time of enrollment and following randomization patients will commence treatment with oral iron. Duration of treatment will be 3 months. Laboratory monitoring will also commence at the time of enrollment along with ongoing evaluation of signs and symptoms of anemia, side effects of oral iron therapy, compliance with oral iron therapy. Duration of monitoring will be 6 months.

A medication diary will be provided to all subjects of each group to track their intake of their oral iron supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Iron Deficiency Anemia
* Pediatric patients (1-18 years of age) without regard of gender, race, ethnicity nor language.
* Able and willing to take oral iron (tablet or liquid).

Exclusion Criteria:

* Pregnant or lactating patients
* Known allergies or intolerance to oral iron formulations
* Concomitant chronic medical conditions affecting iron metabolism
* Short gut syndrome
* Celiac disease
* Inflammatory bowel disease
* Cancer
* Chronic kidney disease
* Blood transfusions in the past 3 months
* IV iron administration in the past 3 months
* Oral iron supplementation in the past 2 weeks

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin stabilization | Change between baseline and 3 months post-enrollment
  Hemoglobin status will be assessed per blood draw at baseline and again at 3 months post-enrollment. Subject will be considered stabilized if hemoglobin levels are within normal range for subject age or demonstrate significant improvement since baseline during that timeframe.
Serum Ferritin stabilization | Change between baseline and 3 months post-enrollment
  Serum Ferritin status will be assessed per blood draw at baseline and again at 3 months post-enrollment. Subject will be considered stabilized if Serum Ferritin levels are within normal range for subject age or demonstrate significant improvement since baseline during that timeframe.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Kheradpour, MD, Principal Investigator — Loma Linda Univeristy

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers. Only study results will be shared.